CLINICAL TRIAL: NCT00928772
Title: The Effect of Cranial Electro Therapy Stimulation in Reducing Perioperative Anxiety for Patients Undergoing First Eye Cataract Surgery
Brief Title: Cranial Electro Therapy Stimulation in Reducing Perioperative Anxiety
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14694
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Anxiety
Keywords: Cranial Electro Stimulation; First Eye Cataract Surgery; Preoperative sedation; Perioperative sedation
MeSH Terms: conditions — Anxiety Disorders | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alpha-Stim intervention (Active Comparator): One hour Alpha-Stim intervention with sham midazolam
  Interventions: Device: CRANIAL ELECTROTHERAPY (Alpha Stim) + SHAM MIDAZOLAM
- Sham Alpha-Stim with midazolam (Sham Comparator): Sham Alpha-Stim intervention with real midazolam administration
  Interventions: Drug: MIDAZOLAM + SHAM ELECTRODES SIMULATING CRANIAL ELECTROTHERAPY
- Placebo (Placebo Comparator): No Alpha-Stim and only topical anesthetics
  Interventions: Other: NO SEDATION WITH SHAM CRANIAL ELECTROSTIMULATION AND PLACEBO VERSED

INTERVENTIONS:
Device: CRANIAL ELECTROTHERAPY (Alpha Stim) + SHAM MIDAZOLAM — APPLYING OF ELECTRODES ON THE EAR LOBES AND TEMPLES WHICH ARE SENDING AN ACTIVE MICROCURRENT THROUGH THE MIDBRAIN PRODUCING SEDATION WITHOUT PHARMACOLOGICAL AGENTS AND GIVING NORMAL SALINE AS A SHAM DRUG SEDATION
  Other Names: AlphaStim
  Arms: Alpha-Stim intervention
Drug: MIDAZOLAM + SHAM ELECTRODES SIMULATING CRANIAL ELECTROTHERAPY — CONVENTIONAL METHOD OF PERIOPERATIVE SEDATION
  Other Names: VERSED
  Arms: Sham Alpha-Stim with midazolam
Other: NO SEDATION WITH SHAM CRANIAL ELECTROSTIMULATION AND PLACEBO VERSED — NO ACTIVE SEDATION, ONLY SHAM ELECTRODES AND NORMAL SALINE SIMULATING MIDAZOLAM.
  Arms: Placebo

SUMMARY:
Cranial electro stimulation (CES) provides safe, adequate, side-effect free sedation without excessive drowsiness in preoperative settings.

DETAILED DESCRIPTION:
CES Alpha-Stim is a non-invasive device which has been in place and has been approved for patients to reduce anxiety by the FDA. This study involves the use of CES Alpha-Stim device applied to the patient 30 minutes before and through-out cataract surgery procedure and then to measure the level of anxiety and discomfort by using a visual analog scale (VAS). We propose that by applying the device the patients will be able to have markedly less level of anxiety and discomfort before and during the surgery and will ultimately avoid the traditional use of sedative or analgesic drugs being used for these kinds of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders between 50 and 90 years old scheduled for an outpatient "first eye" cataract phacoemulsification with topical anesthesia.
* ASA classification I II and III

Exclusion Criteria:

* ASA classification IV (patients with a chronic or severe disease).
* Hypersensitivity to midazolam or benzodiazepines
* acute narrow-angle glaucoma
* untreated open-angle glaucoma
* Patients with any sort of psychiatric or neurological disorder
* Patients on anti-anxiety medication
* Patients who have demand-type pacemakers installed before 1999* *Note: These are the exclusions listed for liability purposes by Alpha-Stim. There are no FDA exclusions.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2009-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grigory Chernyak, Principal Investigator — Oklahoma City VAMC
Locations (1):
- Oklahoma City VA Medical Center, Oklahoma City, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alpha-Stim Intervention | Sham Alpha-Stim With Midazolam | Placebo
Started | 39 | 38 | 38
Completed | 39 | 38 | 38
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alpha-Stim Intervention | Sham Alpha-Stim With Midazolam | Placebo | Total
Number analyzed (Participants) | 39 | 38 | 38 | 115
Age, Customized [Count of Participants; unit: Participants]
  50-90 years | 39 | 38 | 38 | 115
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 39 | 38 | 38 | 115
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 38 | 38 | 115

OUTCOME MEASURES:

1. Primary Outcome: Anxiety During Cataract Surgery Under Topical Anesthesia
Description: Anxiety was accessed via VAS from 0 to 10 with 10 being the most anxious.
Time Frame: during the cataract surgery up to30 minutes
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Alpha-Stim Intervention | Sham Alpha-Stim With Midazolam | Placebo
Number analyzed (Participants) | 39 | 38 | 38
units on a scale | 3.19 [1 to 8] | 2.96 [1 to 9] | 4.10 [1 to 10]

2. Secondary Outcome: Eye Discomfort Perception During Cataract Surgery Under Topical Anesthesia
Description: VAS from 0 to 10 with 10 being maximal discomfort percieved
Time Frame: during cataract surgery up to 30 minutes
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Alpha-Stim Intervention | Sham Alpha-Stim With Midazolam | Placebo
Number analyzed (Participants) | 39 | 38 | 38
units on a scale | 2.58 [1 to 7] | 2.66 [1 to 8] | 2.79 [1 to 8]

3. Secondary Outcome: Mean Arterial Pressure During the Cataract Surgery Under Topical Anesthesia
Time Frame: during cataract surgery up to 30 minutes
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Alpha-Stim Intervention | Sham Alpha-Stim With Midazolam | Placebo
Number analyzed (Participants) | 39 | 38 | 38
mmHg | 99.5 [74.6 to 135.3] | 99.8 [66.7 to 126.3] | 104.5 [79 to 124.5]

4. Secondary Outcome: Heart Rate During Cataract Surgery Under Topical Anesthesia
Time Frame: during cataract surgery up to 30 minutes
Measure: Mean (Full Range); unit: Beats per minute
Arm/Group | Alpha-Stim Intervention | Sham Alpha-Stim With Midazolam | Placebo
Number analyzed (Participants) | 39 | 38 | 38
Beats per minute | 64.6 [53 to 88] | 65.4 [48 to 80] | 67.9 [47 to 98]

ADVERSE EVENTS:
Arm/Group | Alpha-Stim Intervention | Sham Alpha-Stim With Midazolam | Placebo
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 0/39 | 0/38 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No